CLINICAL TRIAL: NCT07171008
Title: The Effect of Ney Music on Pain, Anxiety, Sleep, and Quality of Life in Patients Undergoing Lumbar Disc Surgery
Brief Title: The Effect of Ney Music on Patients Undergoing Lumbar Disc Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Niran Çoban (Other)
Responsible Party: Sponsor-Investigator, Niran Çoban, Asst.Prof., University of Yalova
Organization: University of Yalova (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NS*
Record Dates: First submitted 2025-07-31; First posted 2025-09-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Disc Herniation; Surgery; Nurse's Role
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ney Music (Experimental): Participants in this group will receive a 15-minute ney performance in addition to routine nursing care at specified times before and after lumbar disc surgery. The intervention will be carried out in three sessions:
  I. Session: On the day of surgery, before surgery
  II. Session: Within the first 3 hours after surgery (after transfer to the clinic)
  Session III: Morning of the first day after surgery
  Before and after the application, the Visual Analogue Scale (VAS), State-Trait Anxiety Inventory (STAI-I), Richard-Campbell Sleep Scale, and vital signs (blood pressure, pulse, oxygen saturation) will be measured. Ney pieces in the Rast and Nihavent modes will be used in the sessions.
  Interventions: Other: Ney music
- Standard care (No Intervention): Only standard nursing care will be provided to participants in this group. Parallel to the timing in the intervention group, VAS, STAI-I, Richard-Campbell Sleep Scale, and vital signs will be measured at three separate times (pre-surgery, first 3 hours post-surgery, and first day post-surgery), but no music will be played.

INTERVENTIONS:
Other: Ney music — Ney music concert
  Arms: Ney Music

SUMMARY:
This randomized controlled study aims to investigate the effects of ney music listening, a traditional Turkish wind instrument, on pain, anxiety, sleep quality, and vital signs in patients undergoing lumbar disc herniation surgery. Participants will be randomly assigned to intervention and control groups. The intervention group will receive a 15-minute ney music session at three different time points: preoperative (on the day of surgery), postoperative 3rd hour, and postoperative day 1. The control group will receive standard postoperative nursing care without music intervention. Data will be collected at the same time points in both groups using the Visual Analog Scale (VAS), State-Trait Anxiety Inventory (STAI-I), Richard-Campbell Sleep Questionnaire, and vital signs. The study seeks to evaluate the non-pharmacological benefits of therapeutic music in postoperative recovery.

DETAILED DESCRIPTION:
Lumbar disc herniation is a common spinal disorder that often requires surgical intervention when conservative treatments fail. Although surgery can alleviate nerve compression and reduce pain, many patients continue to experience postoperative pain, anxiety, sleep disturbances, and altered physiological parameters, all of which negatively impact recovery. For this reason, complementary approaches such as therapeutic music have gained attention as supportive strategies in postoperative care.

This randomized controlled trial is designed to evaluate the effect of ney music listening, a traditional Turkish musical practice, on postoperative pain, anxiety, sleep quality, and physiological parameters (heart rate, blood pressure, and oxygen saturation) in patients undergoing lumbar disc surgery. The ney, a reed flute used in classical Turkish music, has been associated with calming and meditative effects, potentially supporting recovery processes.

The intervention group will listen to recorded ney music for 15 minutes in a quiet and dimly lit environment via headphones. The music selection will consist of instrumental compositions in Rast and Nihavend maqams, known for their soothing and relaxing tonalities. Sessions will occur at three specific time points:

Preoperative (the evening before surgery)

Postoperative 3rd hour (after transfer to the clinic)

Postoperative Day 1 (before bedtime)

In each session, pain (measured with the Visual Analog Scale - VAS), anxiety (measured with the State-Trait Anxiety Inventory-I), sleep quality (Richard-Campbell Sleep Questionnaire), and vital signs (systolic and diastolic blood pressure, pulse, and SpO₂) will be assessed before and after music listening in the intervention group.

The control group will receive routine postoperative care without any music intervention. However, outcome measurements will be collected at the same intervals and using the same tools to enable comparison.

The study hypothesizes that listening to ney music may serve as an effective, non-pharmacological method to enhance postoperative comfort by reducing pain and anxiety, stabilizing physiological parameters, and improving sleep quality. The results are expected to contribute to the growing body of evidence supporting the integration of music therapy into clinical nursing practice, particularly in surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone lumbar disc surgery under general anesthesia

  * 18 years old and over,
  * At least 3 hours have passed from the analgesic administration,
  * Patients willing to participate in the study will be included in the study.

Exclusion Criteria:

* Patient-controlled analgesia (PCA) is applied,

  * Over 70 years old,
  * Using anxiolytic and sedative drugs,
  * Having a psychiatric illness,
  * Patients with communication barriers will not be included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The Effect of Ney Music on Pain | 6 month
  Visual Analog Scale: The Visual Analog Scale is a commonly used unidimensional measure for assessing pain intensity. The VAS is a measurement tool ranging from 0 to 10 cm (0 to 100 mm) in length. Since the aim of the study is to determine the effect of the non-pharmacological method used on the current pain, the VAS will be used in the assessment of pain before and after application.
  Measurements will be taken at the following intervals:
  On the day of surgery, before surgery
  Three hours after surgery (after transfer to the clinic)
  On the morning of the first day after surgery
The Effect Ney Music on Anxiety | 6 month
  State Anxiety Inventory: In our study, the State Anxiety Inventory will be used before and after the procedure to assess patients' anxiety levels in a specific situation. The State Anxiety Inventory (STAI-I) is a tool that measures how an individual feels at a specific moment and in a specific situation, i.e., their anxiety level in that situation.Each subscale consists of 20 items, and the inventory consists of a total of 40 items. When calculating the State Anxiety Inventory, the scoring is reversed for items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The total score from both scales in the inventory ranges from 20 to 80. High scores on the scales indicate high anxiety, while low scores indicate low anxiety levels. Measurements will be taken at the following intervals:
  On the day of surgery, before surgery;Three hours after surgery (after transfer to the clinic); On the morning of the first day after surgery
The Effect Ney Music on Sleep | 6 month
  Richard-Campbell Sleep Scale: Assesses the depth of nighttime sleep, the time it takes to fall asleep, the frequency of waking up, the time spent awake after waking up, the quality of sleep, and the noise level in the environment. Each item is rated on a scale ranging from 0 to 100 using the Visual Analog Scale technique. A score between "0-25" on the scale indicates very poor sleep, while a score between "76-100" indicates very good sleep. The total scale score is evaluated based on five items, excluding the 6th item, which assesses the noise level in the environment, with a total score of 22. As the scale score increases, patients' sleep quality also improves.
  It will be used to evaluate the effect of non-pharmacological interventions on patients' sleep levels after surgery.
  Measurements will be taken at the following intervals:
  On the day of surgery, before surgery
  Three hours after surgery (after transfer to the clinic)
  On the morning of the first day after surgery
The Effect Ney Music on blood pressure | 6 month
  Patients' blood pressure, values will be recorded. The effect of non-pharmacological interventions on patients' blood pressure values will be evaluated.
  Measurements will be taken at the following intervals:
  On the day of surgery, before surgery
  Three hours after surgery (after transfer to the clinic)
  On the morning of the first day after surgery
The Effect Ney Music on pulse | 6 month
  Patients' pulse , values will be recorded. The effect of non-pharmacological interventions on patients' pulse values will be evaluated.
  Measurements will be taken at the following intervals:
  On the day of surgery, before surgery
  Three hours after surgery (after transfer to the clinic)
  On the morning of the first day after surgery
The Effect Ney Music on oxygen saturation | 6 month
  Patients' oxygen saturation , values will be recorded. The effect of non-pharmacological interventions on patients' oxygen saturation values will be evaluated.
  Measurements will be taken at the following intervals:
  On the day of surgery, before surgery
  Three hours after surgery (after transfer to the clinic)
  On the morning of the first day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: NİRAN ÇOBAN, Study Director — University of Yalova
Locations (1):
- Niran Çoban, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gezginci E, Iyigun E, Kibar Y, Bedir S. Three Distraction Methods for Pain Reduction During Cystoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain, Anxiety, and Satisfaction. J Endourol. 2018 Nov;32(11):1078-1084. doi: 10.1089/end.2018.0491. PMID 30280915
- [Background] Erdal, B., Kındap Tepe, Y., Öztürk, O. M., Çiğdem, B., Erol, T., Bulut, M. H., et al. (2022). Tarihi Türk müziği makamlarının fizyolojik ve psikolojik etkileri üzerine bir araştırma. Türk Dünyası Sosyal Bilimler Sempozyumu Tam Metin Kitabı. İzmir.
- [Background] Doğan, H. D. (2022). Klasik Türk müziği makamları uygulanarak yapılan hemşirelik doktora tezlerinin değişkenler açısından sistematik incelenmesi. Mersin Üniversitesi Tıp Fakültesi Lokman Hekim Tıp Tarihi ve Folklorik Tıp Dergisi, 12(3), 610-627.
- [Background] Gezginci E, Iyigun E, Yalcin S, Bedir S, Ozgok IY. Comparison of Two Different Distraction Methods Affecting the Level of Pain and Anxiety during Extracorporeal Shock Wave Lithotripsy: A Randomized Controlled Trial. Pain Manag Nurs. 2018 Jun;19(3):295-302. doi: 10.1016/j.pmn.2017.09.005. Epub 2017 Dec 14. PMID 29248604
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Karaman, Ö. Z., Özer, N. (2015). Richard-Campbell Uyku Ölçeği geçerlik ve güvenilirlik çalışması. Türk Uyku Tıbbi Dergisi, 2, 29-32.
- [Background] Leonard H. Live Music Therapy During Rehabilitation After Total Knee Arthroplasty: A Randomized Controlled Trial. J Music Ther. 2019 Feb 16;56(1):61-89. doi: 10.1093/jmt/thy022. PMID 30770536
- [Background] Lin LW, Weng SC, Wu HS, Tsai LJ, Lin YL, Yeh SH. The Effects of White Noise on Agitated Behaviors, Mental Status, and Activities of Daily Living in Older Adults With Dementia. J Nurs Res. 2018 Feb;26(1):2-9. doi: 10.1097/JNR.0000000000000211. PMID 29315202
- [Background] Öner, N., Le Compte, A., Durumluk Sürekli Kaygı Envanteri El Kitabı, 2. Baskı, Boğaziçi Üniversitesi Yayınları, No:333,19.
- [Background] Simcock XC, Yoon RS, Chalmers P, Geller JA, Kiernan HA, Macaulay W. Intraoperative music reduces perceived pain after total knee arthroplasty: a blinded, prospective, randomized, placebo-controlled clinical trial. J Knee Surg. 2008 Oct;21(4):275-8. doi: 10.1055/s-0030-1247831. PMID 18979928